CLINICAL TRIAL: NCT07290842
Title: The Effects of Dietary Nitrate in Patients With Hypertensive Kidney Injury
Acronym: DINO-CKD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gødstrup Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KTM-1-2025
Record Dates: First submitted 2025-11-18; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Hypertension; CKD - Chronic Kidney Disease
Keywords: nitrate; hypertension; beetroot
MeSH Terms: conditions — Hypertension; Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beetroot juice (active) (Active Comparator): nitrate content: 400 mg
  Interventions: Dietary Supplement: Beetroot Juice - Active
- Beetroot juice (placebo) (Placebo Comparator): nitrate free
  Interventions: Dietary Supplement: Beetroot juice placebo

INTERVENTIONS:
Dietary Supplement: Beetroot Juice - Active — Intervention is beetroot juice ("Beet It concentrated beetroot juice shots", James White Drinks Ltd, Ipswich, England) The nitrate content of the juice is standardized. The dose of nitrate will be 70 ml/day corresponding to intake of 6.5 mmol/400 mg of nitrate.
  Arms: Beetroot juice (active)
Dietary Supplement: Beetroot juice placebo — The placebo beetroot juice is a corresponding nitrate free beetroot juice, obtained from the manufacturer ("Beet It nitrate depleted shots", James White Drinks Ltd, Ipswich, England.).
  The placebo juice appears identical to the nitrate containing juice regarding color and taste.
  Arms: Beetroot juice (placebo)

SUMMARY:
The study aims to study the effects of diatery nitrate in patients with hypertension and hypertensive kidney injury.

The study is a randomized, placebo-controlled, double-blinded crossover trial. 14-20 patients with hypertension and CKD I-III will be randomized to receive either nitrate or placebo delivered in the form of beetroot juice.

Effect variables will be measured before and after a 2 week treatment. After a washout period of 14 days, the subjects are crossed over to the opposite treatment.

The study is terminated by measuring effect variables after the second treatment period.

DETAILED DESCRIPTION:
AIM: We aim to investigate the mechanisms behind the cardiovascular and renal effect of nitrates in patients with hypertension and hypertensive kidney injury.

HYPOTHESIS: Dietary nitrate decreases BP and increases renal blood flow. This is independent of renal function or enhanced during low eGFR due to reduced renal clearance of nitrate.

METHODS: The study is a randomized, placebo-controlled, double-blinded crossover trial. 14-20 patients with hypertension and CKD I-III will be randomized to receive either nitrate or placebo delivered in the form of beetroot juice.

Effect variables will be measured before and after a 2 week treatment. After each treatment period effect variables will be measured, including include 24 hour bloodpressure measurment. Technetium(Tc)99m - Diethylenetriamine pentaacetate (DTPA) clearance and water based positron emission tomography computed tomography (PET/CT) is performed only after the intervention periods.

After a washout period of 14 days, the subjects are crossed over to the opposite treatment. The study is terminated by measuring effect variables after the second treatment period.

PERSPECTIVE: The knowledge gained from these studies can lead to improved dietary counselling, which is a promising approach in the treatment of hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Hypertension, treated with a maximum of 2 antihypertensive drugs and unattended office BP < 150/95 mmHg at the screening visit, or newly diagnosed without antihypertensive treatment by 24-hour BP or home BP measurement (above 130/80 or 135/85 respectively), and unattended office BP < 160/100 mmHg.

  * CKD I-III based on hypertensive kidney injury. Patients, who previously met the criteria for CKD I within the last 5 years, but no longer has proteinuria after relevant treatment, can also be included. Diagnosis of CKD I can be based on eGFR and either urine albumin/creatine ration or urine-dipstick test with presence of protein.
  * Albumin/creatinine ratio < 500 mg/g
  * eGFR > 30 ml/min/1,73m2
  * Body Mass Index (BMI) ≤ 35 kg/m2
  * Able to adhere to dietary regimen
  * Fertile women must use safe contraception (oral contraceptive pill, hormonal or copper intrauterine device, vaginal ring, contraceptive implant, transdermal contraceptive patch or contraceptive injections) or abstinence. Excluded from this are postmenopausal woman without menstrual bleeding for at least 12 months before inclusion, surgically sterilized women and women with surgically sterilized partner.

Exclusion Criteria:

* • Diagnosis of heart failure, NYHA II-IV

  * Diagnosis of liver failure
  * Diabetes mellitus (all types)
  * Current malignant disease (other than non-melanoma skin cancer)
  * Indicators of other aetiologies of CKD than hypertensive kidney injury, e.g. through kidney biopsy or biochemistry.
  * Previous kidney transplant recipient
  * History of stroke or transient cerebral ischemic attack
  * Current indication of untreated cardiovascular disease, e.g. planned work-up for ischemia.
  * History of myocardial infarction, apart from non-STEMI more than 1 year prior to the study, if the subject is currently revascularized and relevantly medicated.

Organic nitrate treatment Diagnosed secondary hypertension other than renal parenchymal hypertension (i.e. renal artery stenosis, primary hyperaldosteronism, low renin hypertension etc.)

* Pregnancy or lactation
* Alcohol abuse (intake above the recommended guidelines from Danish Health Authorities)
* Conditions treated with medication that investigator finds may interfere with the effect parameters, and cannot be discontinued during the trial (e.g. atrial fibrillation treated with betablockers)
* If, according to the investigator's assessment, the participant is considered unsuitable to participate.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Changes in 24 h systolic blood pressure | Measured on day 1 and day 15 of the intervention period (This represents baseline and after conclusion of each intervention period)
  Measured by Mobiograph

SECONDARY OUTCOMES:
Diastolic blood pressure | Measured on day 1 and day 15 of the intervention period (This represents baseline and after conclusion of each intervention period)
  Mobil graph with 24 h measurments
Heart rate | Measured on 1 and day 15 of the intervention period (This represents baseline and after conclusion of each intervention period)
  Mobil graph with 24 h measurment
Pulsewave velocity | Measured on day 1 and day 15 of the intervention period (This represents baseline and after conclusion of each intervention period)
  Mobil graph with 24 h measurment
Augmentation index | Measured on day 1 and day 15 of the intervention period (This represents baseline and after conclusion of each intervention period)
  Mobilograph with 24 h measurment
Vascular resistance | Measured on day 1 and day 15 of the intervention period (This represents baseline and after conclusion of each intervention period)
  Mobilograph 24 hour measurments
Reflection index | Measured on day 1 and day 15 of the intervention period (This represents baseline and after conclusion of each intervention period)
  Mobilograph 24 hour measuments
Dipping status | Measured on day 1 and day 15 of the intervention period (This represents baseline and after conclusion of each intervention period)
  Mobilograph 24 hour measurments
Blood pressure variability | Measured on day 1 and day 15 of the intervention period (This represents baseline and after conclusion of each intervention period)
  Mobil graph with 24 h measurment
Unattended office blood pressure | Measured on day 1 and day 15 of the intervention period (This represents baseline and after conclusion of each intervention period)
  Measured on the examination days after 5 minutes rest 3 times by an autoumated ossilometric device in an undisturbed room. The mean of the tre measurments is used.
Renal Blood Flow (RBF) | Measured on Day 15 of each intervention period
  Change in RBF determined by water based PET/CT scans
GFR | Measured on Day 15 of each intervention period
  Change in GFR measured by Tc99m-DTPA clearance
Urine concentration of renal tubular transport proteins | Measured on day 1 and day 15 of the intervention period (This represents baseline and after conclusion of each intervention period)
  Urine excretions of aquaporin 2 (AQP2), thiazide-sensitive sodium-chloride cotransporter (NCC) and distal epithelial sodium channel (ENaC)
Vasoactive hormones | Measured on day 1 and day 15 of the intervention period (This represents baseline and after conclusion of each intervention period)
  Change in plasma levels of aldosterone, renin, brain natriuretic peptide (BNP), atrial natriuretic peptide (ANP), copeptin
Measurements of the NO-system | Measured on day 1 and day 15 of the intervention period (This represents baseline and after conclusion of each intervention period)
  Blood and urine levels of: Nitrite, nitrate, cyclic guanosine monophosphate (cGMP)
Plasma and urine levels of sodium, potassium, creatinine, urea, uric acid, albumin and osmolality | Measured on day 1 and day 15 of the intervention period (This represents baseline and after conclusion of each intervention period)
  Measured in blood and urine (24 h collection). Abbsolute and fractional excretions of sodium and potassium and free water clearence will be calculated.
Body composition measurments from bioimpedance spectroscopy | Measured on day 1 and day 15 of the intervention period (This represents baseline and after conclusion of each intervention period)
  Fresenius Body composition monitor is used, which estimates the compartments in the bodycomposition:
  Extracellular Body Water (L), Total Body Water (L), Intracellular Body Water (L), Overhydration (L)
Body weight | Measured on day 1 and day 15 of the intervention period (This represents baseline and after conclusion of the intervention period)
  Patient weight (kg)
Central Blood pressure | Measured on 1 and day 15 of the intervention period (This represents baseline and after conclusion of each intervention period)
  Sphygmocor measurments
Microvascular function | Measured on 1 and day 15 of the intervention period (This represents baseline and after conclusion of each intervention period)
  Laser speckle contrast imaging

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinic in Nephrology and Hypertension, Gødstrup Regional Hospital and Aarhus University, Herning, Denmark

IPD SHARING:
Plan to Share IPD: No